CLINICAL TRIAL: NCT04163926
Title: Optometric Versus Ophthalmic Follow up of Cataract Surgery Patients in Northern Ireland: A Mixed Methods Study
Brief Title: Optometric Follow-up After Cataract Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The RCT part of the study has been stopped. Due to other issues, funding, other trails and policy changes, the rct will not happen. Interviews will continue but RCT part will not.
Sponsor: Queen's University, Belfast (Other)
Collaborators: Belfast Health and Social Care Trust (Other); Southern Health and Social Care Trust (Other Government)
Responsible Party: Principal Investigator, Nathan Congdon, Chief Investigator, Queen's University, Belfast
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: B17/29
Record Dates: First submitted 2019-08-07; First posted 2019-11-15 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Cataract; Age-related Cataract
Keywords: follow up; post surgery; patient satisfaction; optometrist; ophthalmologist; community care
MeSH Terms: conditions — Cataract; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: Randomised control trial (RCT) control versus usual care
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor will not know the study group assignment of participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group - Post op follow up by trained optometrist (Experimental): Intervention group will have cataract follow up conducted by a trained optometrist 4-6 weeks after surgery in community clinic
  Interventions: Procedure: Intervention Group cataract follow up
- Usual care group - Consultant led post op follow up (Active Comparator): Follow-up at 4-6 weeks after surgery led by consultant ophthalmologist
  Interventions: Procedure: Usual Care consultant follow up

INTERVENTIONS:
Procedure: Intervention Group cataract follow up — Intervention group will have cataract follow up conducted by the referring optometrist 4-6 weeks after surgery
  Arms: Intervention group - Post op follow up by trained optometrist
Procedure: Usual Care consultant follow up — Usual care group - Consultant led post op follow up
  Arms: Usual care group - Consultant led post op follow up

SUMMARY:
This study will investigate the effectiveness of an optometric follow up of cataract surgery versus an ophthalmic surgeon follow up. It will investigate patient satisfaction,safety and cost.

DETAILED DESCRIPTION:
The study will be a mixed-methods study, including a randomized controlled trial in which participants are randomized after cataract surgery to follow up to be consultant led follow up or conducted by a trained optometrist 4-6 weeks following surgery. All participants will then return 6 months after surgery for an additional follow-up visit with an ophthalmologist other than the operating surgeon with patient healthcare satisfaction (main outcome), cost-effectiveness and safety outcomes being measured. A subset of patients and local clinicians will also take part in a one-time, individual, semi-structured interview.

This research will test an alternative model of aftercare for cataract surgeries, which may reduce patient waiting time and inconvenience. In turn, this could help improve patient satisfaction and reduce costs for both patients and the National Health Service (NHS).

Participants will be recruited by operating surgeons. The research will take place in the hospital/clinic/optometrists' offices.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cataract surgery in 1st or 2nd eye for age-related cataract, in the Belfast Trust and Southern Trust
* Willing to participate and give informed consent.

Exclusion Criteria:

* Patients judged by operative surgeon to be of high risk of loss of visual acuity in the operative eye (e.g. end stage glaucoma etc.). Note that patients with ocular comorbidity and previous surgery will not be routinely excluded, nor will monocular patients.
* Patients that were not referred by an optometrist.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-02-28 (Estimated); Primary Completion 2022-08-30 (Estimated); Study Completion 2022-09-28 (Estimated)

PRIMARY OUTCOMES:
Patient Satisfaction following different follow up to cataract surgery (Opthalmic led versus optometric follow up) | At 6 months
  Patient satisfaction will be measured using the patient satisfaction questionnaire (PSQ)-18 at 6 months after surgery The scale include values for general satisfaction, technical quality, interpersonal manner, communication, financial aspects, time spent with doctor and accessibility and convenience.
  Each question is scored between 1 - 5. As some questions have reverse scoring (higher values indicate dissatisfaction) scores are reversed so a 5 will show highest satisfaction and 1 show lowest satisfaction.
  Each item within the subscales will be averaged and results will be given for each of the 7 subscales

SECONDARY OUTCOMES:
Cost | At 6 months
  The total cost per patient visit will be determined and compared
Patient safety | At 6 months
  Patient safety outcomes in the operative eye will include:
  loss of visual acuity >=2 lines Intraocular pressure (IOP) rise >=8 millimetres of mercury (mmHg) post-operative complications as documented by the examining ophthalmologist.
Intraocular pressure (IOP) rise | 6 months
  IOP rise will be compared between the 2 groups in mmHg
Visual Acuity | 6 months
  Visual acuity will be compared between the 2 groups
Post operative complications | 6 months
  Post operative complications will be assessed qualitatively. Surgeons at the 6 month follow up will detail if cornea deep and quiet, wound is intact, intraocular lens centred, posterior capsule intact and clear, anterior vitreous quiet, posterior pole and retina remarkable, signs if infection, retained ens matter and other abnormalities recorded by the surgeon.

OTHER OUTCOMES:
Adherence | At 6 months
  How well patients that have had cataract surgery follow advice for at home care (use of post-operative medication, self-report) and attending follow up medical appointments (as per patient records) will also be compared between the two groups.

IPD SHARING:
Plan to Share IPD: No